CLINICAL TRIAL: NCT00004358
Title: Phase II Study of Calcitonin for Tumoral Calcinosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Purpose: Treatment
Other Study IDs: 199/11925; NU-477
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Calcinosis
Keywords: arthritis & connective tissue diseases; rare disease; tumoral calcinosis
MeSH Terms: conditions — Calcinosis; Arthritis; Connective Tissue Diseases; Rare Diseases | interventions — Calcitonin

INTERVENTIONS:
Drug: calcitonin

SUMMARY:
OBJECTIVES: I. Determine whether intermittent, long-term, subcutaneous administration of calcitonin increases phosphaturia, reduces hyperphosphatemia, and increases intact parathyroid hormone levels in patients with tumoral calcinosis.

II. Determine whether calcitonin reduces or prevents tumor recurrence. III. Determine whether hyperphosphatemia abolishes the normal circadian pattern of serum phosphorus.

IV. Determine how repetitive calcitonin administration alters the biochemical markers of bone metabolism in osteopenic patients with tumoral calcinosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients are treated with subcutaneous injections of salmon calcitonin every 3 weeks. Ondansetron premedication and intravenous hydration are also administered.

Patients are followed for disease progression and tumor recurrence.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically confirmed tumoral calcinosis --Prior/Concurrent Therapy-- Prior surgical resection of calcinotic lesion required

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9
Dates: Start 1992-11

CONTACTS AND LOCATIONS:
Overall Officials: Craig B. Langman, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Children's Memorial Hospital, Chicago, Chicago, Illinois, United States